CLINICAL TRIAL: NCT01868399
Title: Pilot Survey of Dengue Fever in Solomon Islands
Status: Completed | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: Ministry of Foreign Affairs, Republic of China, TAIWAN (Unknown); Ministry of Health and Medical Services, Solomon Islands (Other Government); National Referral Hospital (Other Government)
Responsible Party: Principal Investigator, Wen-Ter Lai (20120080), Superintendent, Kaohsiung Medical University Chung-Ho Memorial Hospital
Other Study IDs: KMUH-IRB-20120080
Record Dates: First submitted 2013-05-27; First posted 2013-06-04 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2016-08

CONDITIONS: Arbovirus Infections
Keywords: dengue virus
MeSH Terms: conditions — Arbovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Remaining samples will be provided to the BioBank for the studies of other infectious diseases pathogens.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Suspected dengue fever subjects: No any intervention
- Community Healty Residents: No intervention

SUMMARY:
Since 2009, Kaohsiung Medical University Hospital organized a medical team to provide the medical service for people in Solomon Islands thru Taiwan Health Center at the local. In addition to Malaria and pulmonary tuberculosis, the investigators also found dengue virus, Japanese Encephalitis virus, Chikungunya virus infections and intestinal parasitic infections might be the existing but overlooked and neglected medical issues in Solomon Islands. These infections show similarity in clinical manifestations and usually difficulty in clinical diagnosis, instead these infections rely on the laboratory identification with good laboratory quality and facility.

DETAILED DESCRIPTION:
In this study, the investigators plan to investigate the local people, either from the community or the hospitals, to identify the prevalence and incidence of dengue fever, including laboratory identification of related infections for differential diagnosis, including Japanese Encephalitis virus, Chikungunya virus and intestinal parasitic infections. Intestinal parasite survey has been the routine long-term service offered by the Kaohsiung Medical University Hospital in Solomon Islands. At the same time, the subjects enrolled in this study will also be asked the common medical illness in Solomon Islands (i.e. malaria, pulmonary tuberculosis and metabolic syndrome etc.) in order to delineate the association of dengue fever and these acute and chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer
* reported dengue virus infection volunteer
* people who understand the purpose of the study and agree the to sign the informed consent

Exclusion Criteria:

* people who refuse to join the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Residents of Solomon Islands
  * people who understand the purpose of the study
  * people who agree to sign the informed consent
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2013-03-22; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Dengue fever | at the time of sampling (blood)
  Clinical manifestations, comorbidity and severity

SECONDARY OUTCOMES:
Co-infection and interplay of dengue-like pathogens | within the first 3 months after blood sampling
  Identification and Analysis of dengue-like illness and pathogens to investigate the interplay between these coinfections

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Ter Lai, MD, Study Chair — Kaohsiung Medical University Chung-Ho Memorial Hospital; Jih-Jin Tsai, MD, Ph. D., Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Tropical Medicine center, Kaohsiung City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided